CLINICAL TRIAL: NCT02570386
Title: A Randomized Controlled Trial of Clinical Effectiveness of Freezing All Embryos Followed by Frozen Thawed Embryo Transfer Compared to Fresh Embryo Transfer, in Women Undergoing In-vitro Fertilization Treatment
Brief Title: Clinical Effectiveness of Frozen Thawed Embryo Transfer Compared to Fresh Embryo Transfer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: very slow recruitment
Sponsor: The University of Hong Kong (Other)
Collaborators: Peking University Third Hospital (Other); Nanfang Hospital, Southern Medical University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 15-001
Record Dates: First submitted 2015-09-29; First posted 2015-10-07 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Subfertility
Keywords: In-vitro fertilization; frozen thawed embryo transfer; fresh embryo transfer
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control arm (Active Comparator): Women allocated to the control arm will either undergo fresh embryo transfer at cleavage stage or extended culture and transfer at blastocyst stage according to local policy. A maximum of 2 embryos or blastocysts will be replaced according to the standard protocol under transabdominal ultrasound guidance. Luteal phase support is given according to local protocols.
  Interventions: Procedure: Fresh embryo transfer
- Intervention arm (Active Comparator): Fresh embryo transfer will not be undertaken in this group. Embryos will be frozen by vitrification or slow freezing at cleavage or blastocyst stage according to standard agreed local protocols. Women will be contacted after 4 weeks and arrangements made for frozen embryo transfer.
  Interventions: Procedure: Frozen embryo transfer

INTERVENTIONS:
Procedure: Fresh embryo transfer — Women allocated to the control arm will either undergo embryo transfer at cleavage stage or extended culture and transfer at blastocyst stage according to local policy. A maximum of 2 embryos or blastocysts will be replaced according to the standard protocol under transabdominal ultrasound guidance. Luteal phase support is given according to local protocols.
  Arms: Control arm
Procedure: Frozen embryo transfer — Fresh embryo transfer will not be undertaken. Embryos will be frozen by vitrification or slow freezing at cleavage or blastocyst stage according to standard agreed local protocols. Women will be contacted after 4 weeks and arrangements made for frozen embryo transfer.
  Arms: Intervention arm

SUMMARY:
The objective of the present randomized controlled study is to compare clinical effectiveness and safety of freezing all embryos followed by frozen-thawed embryo transfer (FET) compared to fresh embryo transfer, in women undergoing IVF treatment.

DETAILED DESCRIPTION:
A total of 800 infertile women undergoing IVF treatment will be randomized into one of the following two groups by computer-generated random numbers:

Fresh embryo transfer group: a single fresh embryo transfer FET group: a single FET following freezing of all embryos in the stimulated IVF cycle

All techniques of IVF including ovarian stimulation, harvesting of oocytes, insemination with specially prepared sperm and embryo culture in the laboratory will be according to local protocols. Once the embryos have been cultured up to day 2 or 3, women with 3 or more suitable quality embryos will be randomized to either fresh embryo transfer (control arm) or FET (Intervention arm).

Control arm Women allocated to the control arm will either undergo embryo transfer at cleavage stage or extended culture and transfer at blastocyst stage according to local policy. A maximum of 2 embryos or blastocysts will be replaced according to the standard protocol under transabdominal ultrasound guidance. Luteal phase support is given according to local protocols.

Intervention arm For those allocated to the intervention arm fresh embryo transfer will not be undertaken. Embryos will be frozen by vitrification or slow freezing at cleavage or blastocyst stage according to standard agreed local protocols. Women will be contacted after 4 weeks and arrangements made for frozen embryo transfer.

After at least 4 weeks women will attend the IVF clinic for the transfer of thawed frozen embryos, either in a natural cycle (in ovulatory women who have regular menstrual cycles) or in a hormonally supported cycle using physiological doses of estrogen and progestogens to mimic normal cyclical changes within the endometrium. The choice between replacing frozen-thawed embryos in a natural or hormonally mediated cycle will be a decision driven by the clinical circumstances.

Embryos or blastocysts will be thawed according to local protocols. The transfer is performed by the team clinician with a maximum of 2 embryos or blastocysts being replaced according to the standard protocol under transabdominal ultrasound guidance. Luteal phase support is given at the discretion of the physician.

Follow up strategy:

A pregnancy test will be carried out 2 weeks after embryo transfer in both arms. All women who have a positive pregnancy test 2 weeks after embryo transfer will undergo a transvaginal ultrasound scan to identify the presence and number of a gestation sac with a fetal heart signifying an ongoing pregnancy. Pelvic scan will be repeated at 8 weeks, 12 weeks, 24 weeks and 36 gestation for fetal growth.

Data on all pregnancy outcomes including early pregnancy losses such as miscarriage or ectopic pregnancy will be collected.

In order to achieve consistency with respect to the collection of outcome, standardised case report forms (CRF) will be completed for each woman at each centre. These CRFs will include details on treatment received, pregnancy outcomes, complications in pregnancy, mode of delivery and birth outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Women under 42 years of age
* Presence of at least 3 embryos suitable to freeze on day 2 or 3 following fertilisation based on the centre's criteria
* Written informed consent

Exclusion Criteria:

* Women using donor eggs/donor sperm
* Women undergoing preimplantation genetic diagnosis
* Women with abnormal uterine cavity shown on hysterosalpingogram or saline infusion sonogram
* Women with hydrosalpinges shown on scanning and not corrected treated
* Women with excessive ovarian response at risk of ovarian hyperstimulation where elective freeze is already planned
* Women with serum progesterone level on day of human chorionic gonadotrophin>1.5ng/ml or 5 nmol/L
* Women whose embryos have not survived freeze-thawing in the past
* Fresh transfer is planned e.g. patients with endometriosis or adenomyosis who have received prolonged downregulation
* Only frozen transfer is planned e.g. patients receiving ovarian stimulation regimens which may have adverse impacts on the endometrium

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 138 (Actual)
Dates: Start 2015-10; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Live birth rate | up to 24 weeks
  A baby born alive after 20 weeks gestation

SECONDARY OUTCOMES:
Miscarriage rate | up to 24 weeks
  Miscarriage before 20 weeks gestation
Clinical pregnancy rates | up to 24 weeks
  Presence of at least one gestational sac on ultrasound at 6 weeks
Ovarian hyperstimulation rate | about 1 month
  Ovarian hyperstimulation rate classified according to Royal College of Obstetrics and Gynaecology in the United Kingdom
Failure of embryos to survive after thawing (per embryo thawed) | around 6 months
  More than 50% of cells lysed on thawing
Cumulative live birth within 6 months of ovarian stimulation | up to 24 weeks
  Live birth from the fresh and frozen thawed embryo transfer
Complications of pregnancy | around 1 years
  Complications of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Ernest HY Ng, MD, Principal Investigator — Department of Obstetrics and Gynaecology, The University of Hong Kong
Locations (1):
- Department of Obstetrics and Gynaecology, Hong Kong, Hong Kong, China

REFERENCES:
- [Derived] Zaat T, Zagers M, Mol F, Goddijn M, van Wely M, Mastenbroek S. Fresh versus frozen embryo transfers in assisted reproduction. Cochrane Database Syst Rev. 2021 Feb 4;2(2):CD011184. doi: 10.1002/14651858.CD011184.pub3. PMID 33539543